CLINICAL TRIAL: NCT04312477
Title: The Correlation Within Diarrhea-predominant Irritable Boewl Syndrome(IBS-D) and Intestinal Microbiota Via C1orf106/Cytohesin-1（CYTH-1） /Adenosine Diphosphate-ribosylation Factor 6（ARF6） Signal Pathway and the Intervention Mechanism of Classic Chinese Compound Formula With Clearing Heat and Promoting Dieresis
Brief Title: Efficacy and Safety of Modified Gegen Qinlian Decoction for Diarrhea-predominant Irritable Boewl Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81830018-1
Record Dates: First submitted 2020-01-15; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2019-08

CONDITIONS: Diarrhea-predominant Irritable Boewl Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Modified Gegen Qinlian Decoction, Oral, 7.2g per bag, 2 times / day, 30 minutes before breakfast and dinner
  Interventions: Drug: Modified Gegen Qinlian Decoction
- Control group (Active Comparator): Bifico(Bifidobacterium triple viable capsule), orally，2 capsules/time, 2 days/time.
  Interventions: Drug: Modified Gegen Qinlian Decoction

INTERVENTIONS:
Drug: Modified Gegen Qinlian Decoction — Modified Gegen Qinlian Decoction contains Pueraria lobata 24g, Scutellaria baicalensis 9g, Coptis chinensis 9g, artillery ginger 9g, talc 9g, roasted licorice 6g, and granules are prepared according to 10:1 production process.

SUMMARY:
Diarrhea-predominant irritable boewl syndrome(IBS-D) seriously affect the quality of life in patients. Clinically, it is effective to apply therapeutic method of clearing heat and promoting diuresis to the common syndrome of dampness-heat. Dysbiosis of intestinal microbiota is closely related to the immune imbalance and intestinal mucosal barrier injury. C1orf106/CYTH-1/ARF6 signal pathway, which derive from intestinal micro environment changes,is the mainly cause of intestinal mucosal barrier injury, and this is may be the common pathogenesis of dampness-heat syndrome in IBS-D . Based on the clinic, the project is to study the effect and mechanism of Chinese compound formula of clearing heat and promoting dieresis in modulating intestinal microbiota dysbiosis, repairing intestinal mucosal barrier and reconstructing intestinal microenvironment. With the combination of metagenomics and metabonomics, the study compare the differences of co-metabolites of intestinal microbiota and host within the healthy people, IBS-D patients with dampness-heat syndrome, to explore the relevance between intestinal flora and host co-metabolites. Furthermore, the experimental study is to clarify the drug targets via C1orf106/ CYTH-1/ARF6 signal pathway.Through the study of association between dampness-heat syndrome in IBS-D and intestinal microbiota, it is of important academic significance to reveal the Chinese theory intension of "homotherapy for heteropathy ".

ELIGIBILITY:
Inclusion Criteria:

1. It meets the diagnostic criteria of diarrhea-predominant irritable boewl syndrome and meets the diagnostic criteria for damp-heat syndrome.
2. Age between 18 and 70 years old.
3. Not taking antibiotics, steroids and other hormones, Chinese herbal preparations in the past week (including) Probiotics such as oral and intravenous), microecological preparations or yogurt.
4. The subject informed and voluntarily signed the informed consent form. ;
5. Have a certain reading ability

Exclusion Criteria:

1. Patients with severe organ, liver, kidney and other major organ diseases, hematopoietic system, nervous system or mental illness;
2. combined with other digestive systemic lesions (such as peptic ulcer), or systemic diseases affecting digestive tract motility (eg hyperthyroidism, diabetes);
3. Those who are or need to continue to use drugs that may affect gastrointestinal function (antidiarrheals, antidepressants, anxiolytics, intestinal flora regulators, antibiotics, etc.);
4. Those with a history of allergic reactions to related drugs and a history of severe food allergies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
IBS symptom severity (IBS-SSS)scale | Change from Baseline disease activity at 4weeks
  The IBS-SSS scale is scored from five aspects: the degree of abdominal pain, the frequency of abdominal pain, the degree of bloating, the degree of defecation satisfaction, and the impact on life.Each score is 0-100 points, and the total score is IBS-SSS scores from the degree of abdominal pain, the frequency of abdominal pain, the degree of abdominal distention, the satisfaction of defecation and the impact on life. Each score is 0-100, and the total score is 0-500. The higher the score, the more serious the disease is.
The Clinical Global Impression of severity Scale ( CGI-S) | 4 weeks

SECONDARY OUTCOMES:
Bristol Stool Form Scale | 4 weeks
PRO scale | 4 weeks
The short form 36 (SF-36) health survey questionnaire | 4 weeks
The scores of TCM(Traditional Chinese Medicine) syndrome | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xiyuanhospital, Beijing, Beijing Municipality, China